CLINICAL TRIAL: NCT01650402
Title: Intensive Versus Standard Blood Pressure Lowering to Prevent Functional Decline in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, William B. White, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11-155S-2; 2R01AG022092-06A1 (NIH)
Record Dates: First submitted 2011-12-14; First posted 2012-07-26 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Hypertension, Systolic; Cerebrovascular Disease
Keywords: Hypertension, systolic; Elderly (> or equal to 75 years); Cerebrovascular disease
MeSH Terms: conditions — Isolated Systolic Hypertension; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive (Experimental): Intensive anti-hypertensive therapies using standard blood pressure medications to lower blood pressure to a level less than or equal to 130 mmHg
  Interventions: Other: Anti-hypertensive therapy to SBP 130 mm Hg
- Standard (Active Comparator): Standard anti-hypertensive therapies using standard blood pressure medications to lower blood pressure to a level less than or equal to 145 mmHg
  Interventions: Other: Anti-hypertensive therapy to SBP 145 mm Hg

INTERVENTIONS:
Other: Anti-hypertensive therapy to SBP 130 mm Hg — Anti-hypertensive therapy to achieve 24 hour systolic blood pressure less than or equal to 130 mm Hg
  Arms: Intensive
Other: Anti-hypertensive therapy to SBP 145 mm Hg — Anti-hypertensive therapy to achieve 24 hour systolic blood pressure less than or equal to 145 mm Hg
  Arms: Standard

SUMMARY:
This randomized clinical trial examines if lowering and maintaining 24-hour ambulatory systolic blood pressure to <130 mmHg (intensive control) versus <145 mmHg (standard control) slows/halts the progression of deterioration of mobility and cognitive function linked to white-matter disease (also known as white-matter hyperintensity or WMH) in patients with normal or mildly impaired mobility and cognition in subjects with detectable cerebrovascular disease (>0.5% WMH fraction of intracranial contents). The study patients will be enrolled and randomized to one of two levels of ambulatory blood pressure control (intensive to achieve a goal 24-hour systolic blood pressure of < 130 mmHg or standard to achieve a goal 24-hour systolic blood pressure of < 145 mmHg) for a total of 36 months.

DETAILED DESCRIPTION:
The study patients will be enrolled and randomized to one of two levels of ambulatory BP control (intensive to achieve a goal 24-hour systolic BP of < 130 mmHg or standard to achieve a goal 24-hour systolic BP of < 145 mmHg) for a total of 36 months. Similar antihypertensive regimens will be used in both of the treatment groups. Titration of antihypertensive therapies will be performed at monthly intervals for the first 3 to 6 months post-randomization to achieve goal systolic BP. The primary and secondary outcomes will be evaluated at baseline, and following 18 months and 36 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* 75 years of age or older
* Seated clinic systolic BP >150 mmHg in the untreated state (see criterion D)
* At risk for cerebrovascular disease (history of smoking, dyslipidemia, type 2 diabetes, longstanding hypertension, family history). Patients must have visible (0.5% WMH or more)white-matter hypertensity lesions on screening magnetic resonance imaging
* To achieve success in maintaining a 24-hour systolic BP of <140-145 mmHg in the standard treatment group or a systolic BP <125-130 mmHg in the intensive treatment group, patients will be eligible for inclusion if (1) their clinic systolic BP is 150-170 mmHg, and they are taking 0 to 2 antihypertensives, (2) their systolic BP is >170 mmHg and they are taking 0 to 1 antihypertensives

Exclusion Criteria:

* Uncontrolled diabetes mellitus (HBA1c >10%)
* History of stroke, dementia or clinically impaired gait (Mini-mental status exam score (MMSE) <24, Short Physical Performance Battery for gait (SPPB) < 9,)
* Body Mass Index > 45 kg/m2 and/or arm circumference > 44 cm)
* Poor kidney function (defined as estimated GFR <30 ml/minute)
* Active liver disease or serum transaminases >3 times the upper limit of normal
* Major cardiovascular event (e.g. myocardial infarction) or procedure (e.g. cardiac bypass surgery) in past 3 months; stroke with residual gait abnormality
* Uncompensated congestive heart failure (NYHA class III or IV or documented ejection fraction <30%)
* Chronic atrial fibrillation that disallows ambulatory BP monitoring to be successfully performed
* Medical conditions that limit survival to < 3 years
* Non-dermatologic cancer diagnosed within 2 years
* Organ transplantation requiring anti-rejection drug therapy
* Severe and unexplained weight loss (>15%) in past 6 months
* Medical need to undergo recurrent phlebotomy or blood transfusions
* Current participation in another investigational trial
* Unable to obtain informed consent
* Factors limiting adherence to the interventions
* MRI contraindications (including MRI-incompatible implants, severe claustrophobia).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 199 (Actual)
Dates: Start 2011-12; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B. White, M.D., Principal Investigator — Pat and Jim Calhoun Cardiology Center, University of Connecticut Health Center; Leslie Wolfson, M.D., Principal Investigator — Department of Neurology, University of Connecticut Health Center
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623
- [Derived] White WB, Wakefield DB, Moscufo N, Guttmann CRG, Kaplan RF, Bohannon RW, Fellows D, Hall CB, Wolfson L. Effects of Intensive Versus Standard Ambulatory Blood Pressure Control on Cerebrovascular Outcomes in Older People (INFINITY). Circulation. 2019 Nov 12;140(20):1626-1635. doi: 10.1161/CIRCULATIONAHA.119.041603. Epub 2019 Oct 14. PMID 31607143
- [Derived] White WB, Jalil F, Wakefield DB, Kaplan RF, Bohannon RW, Hall CB, Moscufo N, Fellows D, Guttmann CRG, Wolfson L. Relationships among clinic, home, and ambulatory blood pressures with small vessel disease of the brain and functional status in older people with hypertension. Am Heart J. 2018 Nov;205:21-30. doi: 10.1016/j.ahj.2018.08.002. Epub 2018 Aug 11. PMID 30145340
- [Derived] White WB, Marfatia R, Schmidt J, Wakefield DB, Kaplan RF, Bohannon RW, Hall CB, Guttmann CR, Moscufo N, Fellows D, Wolfson L. INtensive versus standard ambulatory blood pressure lowering to prevent functional DeclINe in the ElderlY (INFINITY). Am Heart J. 2013 Mar;165(3):258-265.e1. doi: 10.1016/j.ahj.2012.11.008. Epub 2013 Jan 5. PMID 23453090

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intensive | Standard
Started | 99 | 100
Completed | 79 | 86
Not Completed | 20 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive | Standard | Total
Number analyzed (Participants) | 99 | 100 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 99 | 100 | 199
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 51 | 108
  Male | 42 | 49 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 85 | 89 | 174
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mobility - Measured by Change in Gait Speed
Description: Change in gait speed (walking 8 meters) in seconds mediated by the accrual of white-matter hyperintensity lesions (WMH/intracranial cavity volume) using MRI and including degeneration of axonal and myelin components of white matter using MRI technology known as diffusion tensor imaging (DTI).
Time Frame: Change from baseline to 36 months
Population: 78 participants from the intensive group and 86 participants from the standard group were included in the mobility analysis because 1 participant from the intensive group did not complete mobility testing
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intensive | Standard
Number analyzed (Participants) | 78 | 86
seconds | 0.4 (2.0) | 0.42 (2.73)

2. Secondary Outcome: Cognitive Function - as Measured by Change in Stroop Test Score
Description: Change in cognitive function as measured by stroop test score: number of correct responses in 45 seconds.
  The score for the Stroop Test is the number of correct responses provided in 45 seconds on each test condition: word reading, color naming, and inhibition. For the inhibition condition, words are written in an incongruous ink color (e.g., the word red written in blue ink) and participants must provide the ink color. Scores range from 0 to no upper limit, with higher scores indicating better performance.
Time Frame: Change from baseline to 36 months
Population: 69 participants from the intensive group and 76 participants from the standard group were included in analysis because 10 participants in the intensive group and 10 participants in the standard group did not complete cognitive testing
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Intensive | Standard
Number analyzed (Participants) | 69 | 76
correct responses | -2.7 (8.0) | -0.8 (6.4)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout a participant's study completion, an average of 36 months
Arm/Group | Intensive | Standard
All-Cause Mortality (participants affected / at risk) | 2/99 | 4/100
Serious Adverse Events (participants affected / at risk) | 33/99 | 36/100
Other Adverse Events (participants affected / at risk) | 86/99 | 70/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive (N=99) | Standard (N=100)
Arrhythmia (Cardiac disorders) | 3 (3) | 4 (4)
Heart failure (Cardiac disorders) | 0 (0) | 2 (2)
Stroke (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 4 (4)
Pacemaker implantation (Cardiac disorders) | 1 (1) | 2 (2)
Presyncope (Cardiac disorders) | 3 (4) | 2 (2)
Heart stent placement (Cardiac disorders) | 0 (0) | 1 (1)
Other cardiac hospitalizations (Cardiac disorders) | 1 (2) | 2 (2)
Hyperglycemia hospitalization (Endocrine disorders) | 0 (0) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 2 (2) | 2 (5)
Gastrointestinal bleed (Gastrointestinal disorders) | 2 (3) | 1 (1)
Cholecystectomy (Gastrointestinal disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 2 (2)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1)
Breast cancer diagnosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (8)
Pulmonary Emboli (Vascular disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Hospitalization for fall (General disorders) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colon cancer diagnosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic cancer diagnosis (Endocrine disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (3)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Hip surgery (Surgical and medical procedures) | 3 (3) | 4 (5)
Knee surgery (Surgical and medical procedures) | 4 (5) | 0 (0)
Subdural hematoma (Vascular disorders) | 1 (1) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hospitalization for pain (General disorders) | 2 (2) | 1 (1)
Hospitalization for fatigue (General disorders) | 0 (0) | 1 (1)
Hospitalization for weakness (General disorders) | 1 (1) | 0 (0)
Abdominoplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (1) | 1 (1)
Ovarian mass removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Back surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Leg amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Thyroid surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Pump placed for incontinence (Surgical and medical procedures) | 1 (1) | 0 (0)
Death due to cancer (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive (N=99) | Standard (N=100)
Fatigue (General disorders) | 5 (5) | 5 (6)
Fall (General disorders) | 30 (40) | 31 (44)
Edema (Vascular disorders) | 22 (22) | 13 (15)
Urinary Tract Infection (Renal and urinary disorders) | 8 (10) | 9 (12)
Dizziness (Nervous system disorders) | 9 (11) | 6 (7)
Lightheadedness (Nervous system disorders) | 12 (16) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT01650402/SAP_000.pdf
  • Study Protocol (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT01650402/Prot_001.pdf